CLINICAL TRIAL: NCT00852475
Title: Comparative Effects of Two Popular Diets in Veterans With the Metabolic Syndrome
Brief Title: Comparative Effects of 2 Diets in Veterans With the Metabolic Syndrome
Acronym: MUFAPUFA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CARA-030-08F; HP-00040456 (Other: Univ. of MD School of Med IRB)
Record Dates: First submitted 2009-02-26; First posted 2009-02-27 (Estimated); Results first posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2016-12

CONDITIONS: Metabolic Syndrome
Keywords: MUFA; PUFA; MOVE! program
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MUFA (Placebo Comparator): Assignment to monounsaturated enriched diet with exercise. This represents the MUFA MOVE! program
  Interventions: Dietary Supplement: MUFA MOVE! (Monounsaturated fatty enriched diet)
- PUFA (Active Comparator): Assignment to polyunsaturated enriched diet with exercise. This represents the PUFA MOVE! program
  Interventions: Dietary Supplement: PUFA MOVE! (Polyunsaturated fatty acid enriched diet)

INTERVENTIONS:
Dietary Supplement: MUFA MOVE! (Monounsaturated fatty enriched diet) — MUFA MOVE!diet and exercise program
  Arms: MUFA
Dietary Supplement: PUFA MOVE! (Polyunsaturated fatty acid enriched diet) — PUFA MOVE! diet and exercise program
  Arms: PUFA

SUMMARY:
The purpose of the study is to examine the effects of 2 commonly used diets, a Mediterranean monounsaturated fatty acid enriched (MUFA) or AHA polyunsaturated (PUFA) enriched diet combined with the VA Managing Overweight/Obesity for Veterans Everywhere (MOVE!) program so as to determine which one is superior in reducing cardiometabolic risk factors associated with Metabolic Syndrome. The risk factors considered include lipids and lipoproteins, inflammatory markers such as CRP and adiponectin, endothelium-dependent flow-mediated vasodilatation (FMD) and the postprandial lipid responses to a meal.

Cardiometabolic risk factors will be determined by measuring several cardiovascular risk associated parameters including:

Biochemical measurements of lipids and inflammatory markers, body composition and VO2max (Specific Objective 1, Descriptive).

Postprandial response to a meal challenge and endothelial vasoreactivity (FMD) assessed by BART (Specific Objective 2, Physiological).

Determination of the effects on postheparin lipases and transfer protein activity, visceral adipose tissue (VAT) and homeostasis model assessment-estimated insulin resistance (HOMA-IR) (Specific Objective 3, Mechanistic)

DETAILED DESCRIPTION:
The Metabolic Syndrome (MetS) is a common problem among Veterans and is associated with a greater likelihood of cardiovascular disease (CVD). The Mediterranean diet is the only popular diet that has been shown to reduce CVD event rates but the extent to which monounsaturated fatty acid (MUFA) or polyunsaturated fatty acid (PUFA) enrichment results in improvement in parameters of MetS is unresolved. Similarly, while low intensity exercise improves the CVD risk factor profile, there have been no comparative investigations comparing MUFA and PUFA enriched diets and exercise in patients with MetS that have extended beyond 1 year. Recently, the VA established the MOVE! program, a national weight management program designed to help Veterans lose weight. Using the VA promoted program, we will perform a systematic evaluation of the effects of dietary fat composition [comparison between MUFA-enriched and PUFA enriched diet] with MOVE!. We hypothesize that a MUFA-enriched diet consisting of antioxidant, lipid reducing and insulin sensitizing properties will be superior to the less palatable PUFA-enriched diet on improving cardiometabolic parameters associated with MetS. Specifically, the MUFA MOVE! program is expected to lead to greater improvements than the PUFA MOVE! program in body composition and aerobic fitness (Specific Aim 1), endothelial dependent flow mediated vasodilatation and the postprandial lipid response to a meal load (Specific Aim 2) and the mechanisms (lipolytic and lipid transfer protein activity, homeostasis model assessment-estimated insulin resistance) responsible for these effects (Specific Aim 3). Collectively, these studies will advance our understanding of mechanisms underlying the differential effects of MUFA and PUFA-enriched dietary regimens on cardiometabolic health and when combined with the MOVE! program, will provide new and useful information to Veterans (and the general public) interested in optimizing their diets for CVD disease prevention and improved vascular health.

ELIGIBILITY:
Inclusion Criteria:

Presence of 3 or more of the following):

* Waist circumference >102 cm in men or >88 cm women
* Treated Hypertension or Untreated Blood pressure >130/85 and < 160/100 mm Hg
* Treated Hyperglycemia or Untreated Fasting blood glucose (FBG) >100 mg/dL (based on 2006 guidelines)
* Treated Hyperlipidemia or Untreated Triglycerides > 150 mg/dL
* HDL-C < 40 mg/dL men < 50 mg/dL women

Exclusion Criteria:

* Decompensated heart failure (NYHA Class IV);
* Severe Pulmonary disease (Unable to walk on a treadmill at 2.5 mph or greater);
* Chronic renal insufficiency (Cr > 2.5 mg/dL)
* Treated diabetes mellitus with FBG > 180 mg/dL or HbA1C >9g %
* Hematologic or malignant disorders
* Treated SBP >160 mmHg and/or DBP > 95 mmHg ;
* Treated TG > 250 mg/dL
* Use of systemic vasodilators (e.g., nitrates)
* Morbid Obesity (BMI > 50 kg/m2)
* Endocrine (thyroid) or metabolic disorders (unless treated and under control)
* Alcohol consumption greater than (2) 4-ounce glasses of table wine, (2) 12-oz bottles of beer or 2 shots of spirits in men or women
* Active IV drug abuse within the past 6 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miller, MD, Principal Investigator — VA Maryland Health Care System, Baltimore
Locations (1):
- VA Maryland Health Care System, Baltimore, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- MUFA: Assignment to monounsaturated enriched diet (in the form of enriched muffins or oils) with exercise. This represents the MUFA MOVE! program
  MUFA MOVE! (Monounsaturated fatty enriched diet): MUFA MOVE! diet and exercise program
- PUFA: Assignment to polyunsaturated enriched diet (in the form of enriched muffins or oils) with exercise. This represents the PUFA MOVE! program
  PUFA MOVE! (Polyunsaturated fatty acid enriched diet): PUFA MOVE! diet and exercise program
Period: Overall Study
Arm/Group | MUFA | PUFA
Started | 26 | 20
Completed | 23 | 16
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MUFA | PUFA | Total
Number analyzed (Participants) | 26 | 20 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 6 | 2 | 8
Gender [Count of Participants; unit: Participants]
  Female | 16 | 12 | 28
  Male | 10 | 8 | 18
Region of Enrollment [Number; unit: participants]
  United States | 26 | 20 | 86

OUTCOME MEASURES:

1. Primary Outcome: Weight Changes in Veterans With MetS.
Time Frame: 6 months from Baseline
Measure: Mean (Standard Error); unit: kg
Arm/Group | MUFA | PUFA
Number analyzed (Participants) | 23 | 16
kg | -2.3 (0.99) | -6.2 (1.2)

2. Secondary Outcome: Endothelium-dependent FMD Assessed by the Brachial Artery Reactivity Test (BART) at Rest .
Description: Ultrasonographic imaging of the brachial artery (BART) was used to assess endothelium-dependent flow-mediated vasodilation (FMD) in participants at rest. To do this,the blood pressure cuff is inflated to 200 mm Hg and kept inflated for 5 minutes. On immediate release of the cuff, the brachial artery was imaged within 1 minute after cuff release.
Time Frame: 6 months from Baseline
Measure: Mean (Standard Error); unit: percentage of change from baseline
Groups:
- MUFA Arm: Assessment of FMD after six months of MUFA enrichment
- PUFA Arm: Assessment of FMD after 6 months of PUFA enrichment
Arm/Group | MUFA Arm | PUFA Arm
Number analyzed (Participants) | 23 | 16
percentage of change from baseline | 0.19 (0.29) | 1.5 (0.38)

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- MUFA: subjects received a diet enriched in MUFA
- PUFA: subjects received a diet enriched in PUFA
Arm/Group | MUFA | PUFA
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/16
Other Adverse Events (participants affected / at risk) | 0/23 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes